CLINICAL TRIAL: NCT06438822
Title: Second-line Treatment of PD-1 and CTLA-4 Blockade Combined With Liposomal Irinotecan Plus Leucovorin and Fluorouracil for Advanced Cholangiocarcinoma: a Single-arm, Prospective Phase II Trial
Brief Title: Cadonilimab Combined With Liposomal Irinotecan Plus Leucovorin and Fluorouracil for Advanced Cholangiocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Dan Cao, Chief physician, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024（791）
Record Dates: First submitted 2024-05-27; First posted 2024-06-03 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2024-05

CONDITIONS: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — irinotecan sucrosofate; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadonilimab+NIFU regimen (Experimental): There will be two cohorts. Cohort 1 includes patients who have failed first-line treatment with gemcitabine-based chemotherapy combined with PD-L1/PD-1 monoclonal antibody immunotherapy. Cohort 2 includes patients who have failed chemotherapy with gemcitabine-based chemotherapy as a first-line treatment and who had not been treated with PD-L1/PD-1 monoclonal antibody immunotherapy.
  Interventions: Combination Product: Cadonilimab Combined With Liposomal Irinotecan Plus Leucovorin and Fluorouracil

INTERVENTIONS:
Combination Product: Cadonilimab Combined With Liposomal Irinotecan Plus Leucovorin and Fluorouracil — cadonilimab at a dosage of 6 mg/kg on day 1 combined with intravenous liposomal irinotecan at a dosage of 70 mg/m2 for 90 min on day 1 plus leucovorin at a dosage of 400 mg/m2 for 30 min on day 1 and fluorouracil at a dosage of 2400 mg/m2 for 46 h every 2 weeks.

SUMMARY:
This study aimed to evaluate the efficacy and safety of the combination of cadonilimab with liposomal irinotecan plus fluorouracil and leucovorin for the treatment of advanced biliary tract cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with pathologically confirmed locally advanced unresectable or metastatic adenocarcinoma of the bile ducts, gallbladder, or cholangiocellular carcinoma, with primary tumors located in the intrahepatic bile ducts, hilar bile ducts, distal bile ducts, or gallbladder;
2. Progression after prior gemcitabine-based systemic chemotherapy and refused or were intolerable to initial treatment with gemcitabine-based chemotherapy regimens;
3. At least one measurable objective lesion of the tumor according to the RECIST version 1.1 criteria, which must have a maximum diameter of ≥1 cm for spiral CT or ≥2 cm for plain CT or MRI; and should be performed within 28 days prior to enrollment;
4. Aged 18 to 75 years old;
5. Eastern Cooperative Oncology Group performance status (ECOG PS) ≤ 1;
6. Life expectancy of greater than 3 months;
7. Must be able to participate the study voluntarily and sign the informed consent document;
8. Adequate organ and bone marrow function as below:

Absolute neutrophil count ≥1.5*109/L , platelet count ≥75*109/L , hemoglobin ≥90g/L; Alanine aminotransferase, and aspartate aminotransferase ≤2.5 × upper limit of normal; Total bilirubin and serum creatinine ≤1.5 × upper limit of normal.

Exclusion Criteria:

1. Disease-free survival within 5 years due to other malignancies (except for adequately treated basal cell carcinoma of the skin and carcinoma in situ of the cervix);
2. Serious or uncontrolled infectious disease (HIV, HBV DNA > 500IU/ml);
3. Severe uncontrolled acute infection (infection causing a fever of 38℃ or higher)；
4. Severe hepatic or renal insufficiency; or recent history of myocardial infarction (within 3 months)；
5. Current or past autoimmune disease and susceptibility to its reoccurrence;
6. Serious or uncontrolled pleural effusion or ascites;
7. Subjects with a history of active tuberculosis infection within 1 year prior to the first administration of study drug. If in the judgment of the investigator, subjects with more than 1 year prior to the first administration of study drug were considered suitable for enrollment; Subjects with a long history of chronic diarrhea or the presence of complete intestinal obstruction;
8. Subjects requiring systemic therapy with corticosteroids (> 10 mg/day prednisone equivalent dose) or other immunosuppressive drugs within 14 days prior to administration of study drug.
9. Combined with other serious medical and surgical conditions that affected organ function;
10. Participated in other clinical trial within 4 weeks;
11. Pregnant or breastfeeding women or subjects of childbearing potential (males or females with less than 1 year of menopause) who were unwilling to use contraception;
12. Subjects with a history of allergic or hypersensitivity reactions to components of the study drug;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
overall response rate (ORR) | Up to 2 years
  The total number of participants in the intention-to-treat (ITT) population who achieve a complete response (CR) or partial response (PR) will be considered valid, and the statistical results were used to calculate the ORR based on imaging (CT/MRI) using the RECIST v1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang H, Li L, Li X, Ma Y, Yang Y, Cao D. Second-line treatment of PD-1 and CTLA-4 blockade combined with liposomal irinotecan plus leucovorin and fluorouracil for advanced cholangiocarcinoma: study protocol of a single-arm, prospective phase II trial. Ther Adv Med Oncol. 2024 Oct 28;16:17588359241292264. doi: 10.1177/17588359241292264. eCollection 2024. PMID 39492841